CLINICAL TRIAL: NCT03851614
Title: Basket Combination Study of Inhibitors of DNA Damage Response, Angiogenesis and Programmed Death Ligand 1 in Patients With Advanced Solid Tumors
Brief Title: Study of DNA Damage, Angiogenesis, and PD-L1 Inhibitors in Advanced Solid Tumors
Acronym: DAPPER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAPPER-001
Record Dates: First submitted 2019-01-31; First posted 2019-02-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Mismatch Repair Proficient Colorectal Cancer; Pancreatic Adenocarcinoma; Leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — durvalumab; olaparib; cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Olaparib (given orally at a dose of 300 mg twice a day) in combination with Durvalumab (given intravenously at a dose of 1500 mg every 4 weeks)
  Interventions: Biological: Durvalumab; Drug: Olaparib
- Cohort B (Experimental): Cediranib (given orally at a dose of 20 mg daily, 5 days on 2 days off) in combination with Durvalumab (given intravenously at a dose of 1500 mg every 4 weeks)
  Interventions: Biological: Durvalumab; Drug: Cediranib

INTERVENTIONS:
Biological: Durvalumab — Durvalumab is a human immunoglobulin G (IgG)1 kappa monoclonal antibody directed against human PD-L1. Durvalumab selectively binds human PD-L1 with high affinity and blocks its ability to bind to PD-1 and cluster of differentiation (CD)80. The fragment crystallizable (Fc) domain of durvalumab contains a triple mutation in the constant domain of the IgG1 heavy chain that reduces binding to the complement component C1q and the Fc gamma receptors responsible for mediating antibody dependent cell mediated cytotoxicity.
  Other Names: Imfinzi
Drug: Olaparib — Olaparib (AZD2281) is a potent oral poly Poly (ADP-ribose) Polymerase (PARP) enzyme inhibitor (PARP-1, -2 and -3) that is being developed as an oral therapy, both as a monotherapy (including maintenance) and for combination with chemotherapy and other anti-cancer agents. Olaparib specifically traps PARP1 and PARP2 enzymes at sites of damaged DNA; the trapped PARP1- or PARP2-DNA complex is cytotoxic and produces clinical response. Although olaparib also binds to PARP3, recent investigations have suggested PARP-3 inhibition does not contribute towards anti-cancer activity.
  Other Names: Lynparza, AZD2281
  Arms: Cohort A
Drug: Cediranib — Cediranib (AZD2171) is a potent oral small molecule Vascular Endothelial Growth Factor (VEGF) receptor tyrosine kinase inhibitor, specifically inhibiting all three VEGF receptors (VEGFR-1, -2 and -3). It has additional inhibitory activity against stem cell factor receptor tyrosine kinase, and less potency against platelet-derived growth factor receptor tyrosine kinases. Cediranib exerts its anti-angiogenic property by competitively inhibiting the ATP binding site on the VEGF receptors.
  Other Names: AZD2171
  Arms: Cohort B

SUMMARY:
This is a phase 2, single-centre, randomized, multi-cohort trial of subjects with advanced Mismatch Repair Proficient Colorectal Cancer (MMRp-CRC), Pancreatic Adenocarcinoma (PA), and Leiomyosarcoma (LMS). Subjects will be stratified based on their primary malignancy and enrolled into one of the following cohorts:

* Cohort A: olaparib and durvalumab.
* Cohort B: cediranib and durvalumab.

Subjects will receive durvalumab through an intravenous line every 4 weeks. If subjects are assigned to the olaparib group, then they will take this pill twice a day continuously. If subjects are assigned to the cediranib group, then they will take this pill once a day for 5 consecutive days, and then have 2 consecutive days off, every week.

Subjects will be enrolled in this trial to evaluate the changes in genomic and immune biomarkers in tumor, peripheral blood and stool samples, in addition to changes in radiomic profiles. About 90 people (45 subjects in each cohort) will be enrolled into this study at the Princess Margaret Cancer Centre.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the changes in genomic and immune biomarkers in tumor, peripheral blood and stool samples, in addition to changes in radiomic profiles, of subjects with advanced Mismatch Repair Proficient Coloretal Cancer (MMRp-CRC), Pancreatic Adenocarcinoma (PA), or Leiomyosarcoma (LMS) during combination treatment of durvalumab (inhibitor of PD-L1) with either olaparib (inhibitor of Poly (ADP-ribose) polymerase [PARP]) or cediranib (inhibitor of Vascular Endothelial Growth Factor Receptor [VEGFR] tyrosine kinases).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥18
* ECOG 0-1
* Have histologically/cytologically-documented, locally-advanced, or metastatic mismatch repair proficient colorectal cancer (MMRp-CRC), pancreatic adenocarcinoma (PA), or leiomyosarcoma (LMS) that is incurable and has either (a) failed prior standard therapy, (b) for which no standard therapy exists, or (c) standard therapy is not considered appropriate by the subject and treating physician
* Allowable: prior immune-oncology therapy, no maximal limit to the number of prior lines of systemic therapy for advanced or metastatic disease. All prior anti-neoplastic systemic therapy, including immune-oncology, must have a 4 week wash out period. There is no limit to the number of prior anti-neoplastic systemic treatments used before trial enrolment
* Must have at least 1 tumor site that is amendable to tumor biopsy
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 4 weeks (28 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided will not be eligible for this study. Subjects who have archival tissue available, not older than 6 months and with no intervening therapies from the day of the biopsy and the initiation of the study, will also be requested to also submit this sample, but are still required to undergo a pre-treatment biopsy.
* Consent to provide archival tumor tissue for correlative biomarker studies
* Must have at least 1 tumor site that is RECISTv1.1 measurable by CT or MRI scan. A previously irradiated lesion can be considered a target lesion if the lesion is well defined, measurable and there is objective evidence of progression following radiotherapy. The biopsy lesion cannot be the same as the target lesion
* Life expectancy ≥ 16 weeks from proposed first dose date
* Female subject of childbearing potential should have two negative pregnancy tests as verified by the investigator prior to starting any investigational product therapy: serum pregnancy test at screening and negative serum or urine pregnancy test on Cycle 1, Day 1 prior to treatment, and confirmed prior to each subsequent cycle of treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. They must agree to pregnancy testing after the last dose of durvalumab, olaparib or cediranib. This applies even if the subject practices complete abstinence from heterosexual contact
* Females of childbearing potential who are sexually active with a non-sterilized male partner must agree to practice true abstinence or at least two effective methods of contraception from 28 days prior to starting durvalumab, olaparib or cediranib, and agree to continue using such precautions while taking durvalumab, olaparib or cediranib and for 90 days following the last dose of investigational product(s). Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. They must also refrain from egg cell donation and breastfeeding during study participation and for at least 90 days after the final dose of investigational product(s)
* Non-sterilized males who are sexually active with a female partner of childbearing potential must agree to use at least two effective methods of contraception from Day 1 through 90 days after receipt of the final dose of investigational product(s). In addition, they must refrain from sperm donation for 90 days after the final dose of investigational product(s). Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Adequately controlled thyroid function, with no symptoms of thyroid dysfunction. Elevated thyroid stimulating hormone (TSH) with normal free T3 and free T4 are allowed; subjects on thyroid replacement therapy are allowed
* Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below. Subjects are not allowed to have received blood transfusion upwards of 28 days prior to study treatment

  2.Cohort A
* Subjects with MMRp-CRC, PA or LMS with the presence or absence of DDR and HRR (homologous recombination repair) genes will be evaluated retrospectively but it is not an eligibility criterion. Prior PARP usage, including olaparib, is excluded, but other DDR pathway inhibitors are allowed

  3. Cohort B
* Prior antiangiogenic treatment is allowed.

Exclusion Criteria:

1. All cohorts

   * Involvement in the planning and/or conduct of the study or previous enrolment in the present study
   * Subjects with another malignancy unless curatively treated with no evidence of disease for ≥ 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ, Stage 1, grade 1 endometrial carcinoma. Patients with a history of localized triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
   * Untreated central nervous system (CNS) metastatic disease, leptomeningeal disease, or cord compression. Subjects with previously treated brain metastases may participate provided they are stable, have no evidence of new or enlarging brain metastases, and are not using steroids for at least 14 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability. Subjects with a history of treated asymptomatic CNS metastases are eligible, provided they meet all of the following criteria:

     * Measurable disease outside the CNS
     * Only supratentorial metastases allowed
     * No history of intracranial hemorrhage
     * No ongoing requirement for corticosteroids as therapy for CNS disease; anticonvulsants at a stable dose allowed
     * No stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to Day 1 of the study
     * No evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
   * Participation in another clinical study with an investigational product during the last 28 days or 5 half-lives prior to study Day 1. Concurrent enrolment in an observational clinical study or the follow-up period of an interventional study is allowed
   * Subjects receiving any systemic chemotherapy, radiotherapy, within 4 weeks from the last dose prior to study treatment.
   * Receiving, or having received during the four weeks prior to study entry, corticosteroids for any reason. The following are exceptions to this criterion:

     * Intranasal, inhaled, topical, or local steroid injections
     * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
     * Steroids as premedication for hypersensitivity reactions
   * Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of investigational products. Vaccination with a killed vaccine is permitted at any time with consultation with the Principal Investigator
   * Major surgery within 28 days prior to Day 1 of the study or still recovering from prior surgery. Local procedures are allowed if completed at least 24 hours prior to the administration of the first dose of study treatment
   * Any unresolved toxicity NCI CTCAE v5.0 Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, hypothyroidism and the laboratory values defined in the inclusion criteria

     * Patients with Grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician
     * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment by the investigation product may be included only after consultation with the Study Physician
   * Any prior unresolved NCI CTCAE v5.0 Grade > 1 irAE while receiving any previous immunotherapy agent with exception of chronic endocrinopathy that is stable on hormone replacement. Subjects who developed Grade 2 or 3 irAE that has since resolved can be discussed with the Principal Investigator.
   * Diagnosis of autoimmune-based rheumatologic disease or clinically significant autoimmune disorders. Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment are not excluded. Subjects with hypothyroidism on thyroid supplements are not excluded
   * History of primary immunodeficiency
   * Previous allogenic bone marrow transplant or double umbilical cord blood transplantation
   * History of hypersensitivity to durvalumab, olaparib, cediranib or any excipient
   * Measurable mean value QTcF > 470 msec on resting triplicate ECG within a 24 hour period, or if resting ECG indicates uncontrolled, potentially reversible cardiac conditions, or patients with congenital or family history of long QT syndrome
   * Subjects with relative hypotension (< 100/60 mm Hg) or clinically relevant orthostatic hypotension, including a fall in blood pressure of > 20mm Hg
   * A history of poorly controlled hypertension or resting blood pressure > 150/100 mmHg in the presence or absence of a stable regimen of anti-hypertensive therapy

     ---Adequately controlled BP: systolic BP ≤ 140 mmHg and diastolic BP ≤ 90 mmHg in the presence or absence of a stable regimen of antihypertensive therapy.
   * Left ventricular ejection fraction < lower limit of normal (LLN) per institutional guidelines, or <55%, if threshold for normal is not otherwise specified by institutional guidelines, for patients with the following risk factors:

     * Prior or planned treatment with anthracyclines
     * Prior treatment with trastuzumab
     * Prior central thoracic radiation therapy (RT), including exposure of heart to therapeutic doses of ionizing RT
     * History of myocardial infarction within 6 to 12 months prior to randomization
     * Prior history of other significant impaired cardiac function
   * Refractory nausea and vomiting, chronic gastrointestinal diseases or previous significant bowel resection that would preclude adequate absorption of oral drugs
   * History of bowel obstruction within 1 month prior to starting study drugs
   * Subjects unable to swallow orally administered medication
   * Subjects may not have current dependency on IV hydration or total parenteral nutrition
   * Subjects with uncontrolled seizures
   * Active infection requiring systemic antibiotics, antifungal or antiviral drugs
   * Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any subject known to have active tuberculosis, hepatitis B, hepatitis C or human immunodeficiency virus, immunocompromised patients, or any patients with a psychiatric disorder that prohibits obtaining informed consent. Subjects who have had adequately treated tuberculosis may be enrolled upon discussion with Principal Investigators. Subjects who have had prior hepatitis B and C and are not carriers, or have been cured with antivirals, are eligible
   * Female subjects who are pregnant, breast-feeding or male or female subjects of reproductive potential who are not employing an effective method of birth control
   * History of myocardial infarction within 6 months prior to registration
   * History of stroke or transient ischemic attack within 6 months prior to registration
   * Heart failure class III or IV
   * Current cardiac arrhythmia requiring concurrent use of anti-arrhythmic drugs
   * History of hypertensive crisis or hypertensive encephalopathy within 3 years prior to registration, or poorly controlled hypertension at time of registration
   * Clinically significant peripheral vascular disease or abdominal aortic aneurysm (> 5 cm) or aortic dissection. If known history of abdominal aortic aneurysm with ≥ 4 cm in diameter, all of the following must be met: an ultrasound within the last 6 months prior to registration will be required to document that it is ≤ 5 cm; subjects must be asymptomatic from the aneurysm; blood pressure must be well controlled as defined in this protocol
   * Unstable angina within 6 months prior to randomization
   * History of hemoptysis or any significant bleeding within the last 1 month prior to enrollment
   * Presence of cavitation of central pulmonary lesion
   * History of abdominal fistula, intra-abdominal abscess, or gastrointestinal perforation, within the 3 months prior to enrollment
   * Subjects may not have history of bleeding diathesis or coagulopathy. Therapeutic anticoagulation for prior thromboembolic events is permitted but must be discussed with the PI. Subjects requiring two or more anti-thrombotic agents, including anti-platelet agents will be excluded
   * Any condition that would interfere with evaluation of study treatment or interpretation of subject safety or study results.
   * Subjects who are involuntarily incarcerated or are unable to willingly provide consent or are unable to comply with the protocol procedures
   * Subjects who require blood transfusion within 28 days prior to study entry to maintain Hgb > 100 g/L or platelets > 100 x 109/L. Whole blood transfusions in the last 120 days prior to entry to the study are acceptable, outside of 28 days prior to treatment
2. Cohort A (olaparib, durvalumab)

   * Concomitant use of known strong CYP3A inhibitors or moderate CYP3A inhibitors. The required washout period prior to starting study treatment is 2 weeks
   * Concomitant use of known strong or moderate CYP3A inducers . The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
   * If clinically indicated, subjects may not have features suggestive of myelodysplastic syndrome or acute myelogenous leukemia on peripheral blood smear or bone marrow biopsy.
3. Cohort B (cediranib, durvalumab)

   * A major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting cediranib
   * Concomitant use of known strong cytochrome (CYP) 3A inhibitors or moderate CYP3A inhibitors. The required washout period prior to starting study treatments is 2 weeks for strong inhibitors, and at least 1 week for moderate inhibitors
   * Concomitant use of known strong CYP3A inducers or moderate CYP3A inducers. The required washout period prior to starting study treatments is 5 weeks for enzalutamide or phenobarbital and 4 weeks for other agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in genomic and immune biomarkers that will be measured in the baseline biopsy and the first on-treatment biopsy by applying a log-transformation and the t-test. | 3 years
  If a departure from the normal distribution will be noticed for the distributions of the CD8 and CD4 then a log-transformation will be applied. The CD8 and CD4 will be compared between responders and non-responders by applying the t-test. Subgroup analysis based on the site will also be attempted.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 3 years
  Overall response rate (ORR)
Clinical benefit rate (CBR) | 3 years
  Clinical benefit rate (CBR)
Progression-free survival (PFS) | 3 years
  Progression-free survival (PFS)
Overall survival (OS) | 3 years
  Overall survival (OS)
Antitumor activity based on iRECIST | 3 years
  Antitumor activity based on iRECIST
Incidence of treatment-emergent adverse events (AEs) | 3 years
  Incidence of treatment-emergent adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No